CLINICAL TRIAL: NCT05679752
Title: Effects of Massage Therapy and Facial PNF in Early Bell's Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neuro Counsel Hospital, Pakistan (Other)
Collaborators: Al Nafees Medical Hospital, Islamabad (Unknown); Reliance Hospital Rawalpindi (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 338
Record Dates: First submitted 2022-12-15; First posted 2023-01-11 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Bell Palsy
MeSH Terms: conditions — Bell Palsy | interventions — Muscle Stretching Exercises; Massage

STUDY DESIGN:
Intervention Model Description: Randomized control trail
Who Masked: Participant
Masking Description: single blind RCT in which just participants do not know in which group they are being treated
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (Active Comparator): massage therapy will be given to this group of participants
  Interventions: Other: Massage therapy
- experimental group (Experimental): Facial PNFtechnique will be given to this group of participants
  Interventions: Other: Facial PNF technique

INTERVENTIONS:
Other: Facial PNF technique — Stimulation techniques used to facilitate the weak muscle groups
  Other Names: Proprioceptive Neuromuscular Facilitation
  Arms: experimental group
Other: Massage therapy — frictional massage to stimulate the weak muscle groups
  Other Names: Passive massage
  Arms: control group

SUMMARY:
Effects of Massage therapy and Facial PNF in early Bell's palsy

DETAILED DESCRIPTION:
It is an interventional study in which investigator will give massage therapy to one group of patients and facial PNF techniques to other group to evaluate the efficacy of these intervention on bell's palsy pateints

ELIGIBILITY:
Inclusion Criteria:

* Both males and females with age between 20 to 50 years
* All patients diagnosed with Bell's palsy
* Non traumatic onset
* Acute onset 1 to 3 weeks
* Either right or left side

Exclusion Criteria:

* Subject who have other Neurological disorder
* Subjects who have impaired cognition
* Complete paralysis of face
* Open wound on face

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2022-12-14 (Actual)

PRIMARY OUTCOMES:
Sunnybrook facial grading scale | assessment will be done after 6 weeks
  complete tool for assessing facial movement outcomes. Lower score (Zero) means complete paralysis and higher (100) means normal
Facial Clinimetric Evaluation Scale | assessment will be done after 6 weeks
  to evaluate the impairment and disability associated with facial weakness. It is calculated ranging from 0 (worst) to 100 (best)

CONTACTS AND LOCATIONS:
Locations (1):
- Al Nafees Medical Hospital, Islamabd, Islamabad, Federally Administered Tribal..., Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
Still not decided about this.